CLINICAL TRIAL: NCT02286037
Title: Delineating Areas of Secondary Hyperalgesia: Influence of the Assessment Method
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Ringsted, Cand. Scient. San., Rigshospitalet, Denmark
Other Study IDs: H1-2013-045
Record Dates: First submitted 2014-02-07; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Measurements of Areas of Secondary Hyperalgesia
Keywords: Secondary Hyperalgesia; Method; Pin-prick; Monofilament
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Assessments of mechanical skin sensitivity include psychophysical responses to stimulation with calibrated polyamide monofilaments.

One of the applications of polyamide monofilaments are the assessments of magnitude of secondary hyperalgesia areas (SHAs), i.e. areas in normal skin near an injury with increased mechanical sensitivity.

The objective of the study is to investigate the hypothesis, based on previous studies, that a light tactile stimulus delineates a larger SHA than stimulation with a more rigid monofilament.

Twenty-three healthy participants were included in this randomized, two-observer, test-retest study.

A highly significant positive correlation between the bending force of the polyamide filaments and the magnitude of SHA was demonstrated. The "weighted-pin" instrument showed significantly and consistently larger areas than the polyamide monofilaments.

The hypothesis was rejected: a light tactile stimulus did not delineate a larger secondary hyperalgesia area than stimulation with a more rigid monofilament. The "weighted-pin" instrument seems an alternative to the conventional polyamide monofilaments.

DETAILED DESCRIPTION:
Introduction Assessments of mechanical skin sensitivity include psychophysical responses to stimulation with calibrated polyamide monofilaments. Although the theoretical background and the application of monofilaments are straightforward, inconsistencies of the method have been reported in the literature. One of the applications of polyamide monofilaments are the assessments of magnitude of secondary hyperalgesia areas (SHAs), i.e. areas in normal skin near an injury with increased mechanical sensitivity. Secondary hyperalgesia is a measure of central sensitization and reflects the effect of an injury on the central nervous system. The objective of the study is to investigate the hypothesis, based on previous studies, that a light tactile stimulus delineates a larger SHA than stimulation with a more rigid monofilament.

Method Twenty-three healthy participants were included in this randomized, two-observer, test-retest study. The volunteers were blinded to the test-results. The design was adjusted to examine intra-/inter-observer and intra-/inter-day variability in SHAs after a first degree burn injury was induced by a contact thermode (47ºC, 7 minutes, thermode area 12.5 cm2) on the lower leg. The SHAs were assessed 45 to 75 min (15 min for each observer) after the burn injury and delineated by 3 different polyamide monofilaments (50, 299, 986 mN) and a "weighted-pin" instrument (512 mN). The testing order of the monofilaments was randomized, and the observers were blinded to the study results of each other. The examination order of the observers on Day 1 was reversed on Day 2 (> 6 weeks later).

ELIGIBILITY:
Inclusion criteria:

* Healthy
* Age ≥18 years and ≤ 35 years
* Written informed consent
* Urine sample without any trace of opioids (morphine, methadone, buprenorphin)
* Body Mass Index: 18 < BMI < 32 kg/cm2

Exclusion criteria:

* Inadequate psychomotor ability to cooperate
* Inability to understand Danish or English
* Participated in another study in the preceding 60 days
* Known neurological disease
* Use of psychoactive drugs (benzodiazepines, SSRI, TCA, SNRI)
* Alcohol or drug abuse
* Chronic pain
* Use of pain medication on a regular basis
* Skin lesions in the examination area
* Use of prescription medicine 1 week before examination
* Use of over-the-counter (OTC) drugs 48 hours before examination
* Smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
comparison of secondary hyperalgesia areas assessed by the polyamide filaments | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Ringsted, Nurse,cand., Principal Investigator — Rigshospitalet, Denmark